CLINICAL TRIAL: NCT00022126
Title: A Study of Modified Augmented BFM Therapy for Infants With Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy With or Without Donor Bone Marrow Transplantation in Treating Infants With Previously Untreated Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AALL01P1; COG-AALL01P1 (Other: Children's Oncology Group); CDR0000068787 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; acute undifferentiated leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Asparaginase; Cyclophosphamide; Cyclosporine; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Mercaptopurine; Methotrexate; Methylprednisolone; pegaspargase; Thioguanine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Modified Augmented BFM Therapy (Experimental)
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cyclosporine; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: mercaptopurine; Drug: methotrexate; Drug: methylprednisolone; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate; Procedure: allogeneic bone marrow transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: mercaptopurine
Drug: methotrexate
Drug: methylprednisolone
Drug: pegaspargase
Drug: thioguanine
Drug: vincristine sulfate
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Giving the drugs in different combinations may kill more cancer cells. Bone marrow transplantation allows the doctor to give higher doses of chemotherapy and kill more cancer cells.

PURPOSE: Phase II trial to compare the effectiveness of combination chemotherapy with or without donor bone marrow transplantation in treating infants who have previously untreated acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of dexamethasone-based induction chemotherapy followed by augmented Berlin-Frankfurt-Munster (BFM) consolidation chemotherapy with or without allogeneic bone marrow transplantation in infants with previously untreated acute lymphoblastic leukemia.
* Determine the event-free survival of patients treated with this regimen.
* Determine the clinical prognostic features associated with outcome in these patients.
* Compare the biologic characteristics of the leukemia cells with outcome in these patients.

OUTLINE: This is a multicenter study.

Patients receive induction therapy comprising oral dexamethasone 3 times daily on days 1-14; daunorubicin IV on days 1, 8, and 15; vincristine IV on days 1, 8, 15, and 22; and asparaginase intramuscularly (IM) on days 4, 6, 8, 11, 13, 15, 18, 20, and 22. Patients also receive methotrexate intrathecally (IT) on days 1, 8, and 15 (and days 4 and 22 for overt CNS disease).

Patients with M1 or M2 marrow after induction therapy receive augmented consolidation therapy when blood counts recover. Patients receive cyclophosphamide IV on days 1 and 29; cytarabine IV or subcutaneously (SC) on days 2-5, 9-12, 30-33, and 37-40; oral mercaptopurine on days 1-14 and 29-42; vincristine IV on days 15, 22, 43, and 50; pegaspargase IM on days 15 and 43; and methotrexate IT on days 1, 8, and 15.

Patients who do not receive bone marrow transplantation (BMT) proceed to interim maintenance #1 when blood counts recover. Patients receive methotrexate IT on days 1, 11, 22, and 32; methotrexate IV and vincristine IV on days 1, 11, 22, 32, and 43; and pegaspargase IM on days 2 and 23.

When blood counts recover, patients receive delayed intensification #1 comprising vincristine IV on days 1, 8, 15, 43, and 50; doxorubicin IV on days 1, 8, and 15; oral dexamethasone 3 times daily on days 1-7 and 15-21; pegaspargase IM on days 4 and 43; cyclophosphamide IV on day 29; methotrexate IT on days 29 and 36; oral thioguanine on days 29-42; and cytarabine IV or SC on days 30-33 and 37-40.

When blood counts recover, patients receive interim maintenance #2 comprising vincristine as in interim maintenance #1; methotrexate IT on day 1 and IV on days 1, 11, 22, 32, and 41; and pegaspargase IM on days 2 and 23.

When blood counts recover, patients receive delayed intensification #2 comprising vincristine, doxorubicin, dexamethasone, pegaspargase, cyclophosphamide, cytarabine, and thioguanine as in intensification #1. Patients also receive methotrexate IT on days 1 and 29.

When blood counts recover, patients receive maintenance therapy comprising methotrexate IT on day 1 and orally on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; vincristine IV on days 1, 29, and 57; oral dexamethasone 3 times daily on days 1-5, 29-33, and 57-61; and oral mercaptopurine daily. Treatment repeats every 84 days for 6 courses.

Patients with an allergy to pegaspargase replace it with asparaginase IM on the days after receiving methotrexate IV during interim maintenance #1 and #2 and daily over 6 days in place of each dose of pegaspargase during delayed intensification #1 and #2.

After augmented consolidation therapy, patients meeting the following criteria may receive BMT in place of chemotherapy:

* In remission
* Exhibiting chromosome translocation involving 11q23 or Ph+{(9;22)}
* Available HLA-A, B, DR genotypic identical relative donor
* No uncontrolled infection
* Adequate organ function Within 3-4 weeks of consolidation therapy, patients undergoing allogeneic BMT receive cytarabine IV over 1 hour on days -8 to -5; cyclophosphamide IV over 30 minutes on days -7 and -6; and methylprednisolone IV twice daily on days -2 to 0. Patients also undergo total body irradiation twice daily on days -3 to 0. Patients receive allogeneic BMT on day 0. Patients also receive cyclosporine IV every 12 hours beginning on day -1, switching to oral when possible, and continuing until day 60. Patients then taper cyclosporine over the next 60-120 days.

Patients are followed every 2 months for 1 year, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1-2 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 20-40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of previously untreated acute lymphoblastic leukemia (ALL) or acute undifferentiated leukemia

  * CNS or testicular disease allowed
* No L3 sIg+ ALL or acute myelogenous leukemia
* At least 36 weeks gestation for congenital ALL

PATIENT CHARACTERISTICS:

Age:

* Under 366 days at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Steroid therapy within 48 hours of study allowed if complete blood counts and lumbar puncture results known
* No chronic steroid treatment for other disease

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent cytotoxic therapy

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2002-11; Primary Completion 2005-01 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Establish whether the CCG Augmented Regimen (AR) can be successfully administered in the infant age group

SECONDARY OUTCOMES:
Grade 3 or 4 non-hematologic toxicity rates
Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Gaynon, MD, Study Chair — Children's Hospital Los Angeles
Locations (51):
- United States (47):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital of Denver, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Children's Hospitals and Clinics - Minnesota, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Cancer Center, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Australia (2):
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia